CLINICAL TRIAL: NCT04234646
Title: Patient Navigation 2.0: Addressing the Challenge of Scaling Navigation Through Checklist-based Implementation
Brief Title: Patient Navigation 2.0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northeastern Illinois University (Other)
Responsible Party: Principal Investigator, Melissa Simon, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00211685
Record Dates: First submitted 2020-01-14; First posted 2020-01-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: One-on-One Patient Navigation (Active Comparator): One-on-one Patient Navigation will be based on a Case Management Model where patients navigators perform appointment scheduling and reminders; facilitate communication between patients and care teams; and identify and reduce patient barriers through education, outreach, and referrals to community, local, and state resources.
  Interventions: Behavioral: One-on-one Patient Navigation (PN)
- Group 2: Patient Navigation 2.0 Checklist (Experimental): The PN 2.0 Checklist intervention is centered on a learning health system checklist that enumerates a patient's Social Determinants of Health (SDoH) related barriers and tracks completion of services to address SDoH (at community oncology and community social service settings) as well as completion of USPSTF recommended cancer-related screenings, behavioral counseling, and immunizations.
  Interventions: Behavioral: Patient Navigation (PN) 2.0 Checklist

INTERVENTIONS:
Behavioral: Patient Navigation (PN) 2.0 Checklist — The PN 2.0 Checklist intervention is centered on a learning health system checklist that enumerates a patient's Social Determinants of Health (SDoH) related barriers and tracks completion of services to address SDoH (at community oncology and community social service settings) as well as completion of USPSTF recommended cancer-related screenings, behavioral counseling, and immunizations.
  Arms: Group 2: Patient Navigation 2.0 Checklist
Behavioral: One-on-one Patient Navigation (PN) — The one-on-one Patient Navigation will be based on a Case Management Model where PNs perform appointment scheduling and reminders; facilitate communication between patients and care teams; and identify and reduce patient barriers through education, outreach, and referrals to community, local, and state resources
  Arms: Group 1: One-on-One Patient Navigation

SUMMARY:
This study evaluates whether a "Patient Navigation 2.0 Checklist" intervention is effective in addressing patients' social determinants of health and recommended cancer-related screenings, behavioral counseling, and immunizations.

DETAILED DESCRIPTION:
Cancer patient navigation (PN) is an effective strategy for resolving patient barriers to care and improving completion and consistency of cancer screening, follow-up of abnormal findings, and treatment initiation. However, as the current standard one-on-one PN model is challenging to scale across cancers and economically difficult to sustain, the investigators propose to convert one-on-one PN into a learning health system "PN 2.0 Checklist" that will help coordinate navigation workflow and integrate clinical team members with community/local resources. This pragmatic, randomized trial tests whether this checklist strategy is as effective as one-on-one PN in addressing patients' social determinants of health and recommended cancer-related screenings, behavioral counseling, and immunizations.

In this study, half of the participants will be navigated using the "PN 2.0 Checklist". The other half will be navigated using the "One-on-One PN". All participants enrolled in the study will be asked to report their utilization of health services and be asked to complete a patient survey at the beginning of the program and every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Reside in one of the eight Chicago zip codes corresponding to Chinatown's geographical boundaries: 60605, 60607, 60608, 60609, 60616, 60623, 60632, 60653
* Self-identify as Chinese
* Not cognitively impaired
* Have the ability to participate in verbal survey in Cantonese, English, Mandarin, or Toishanese

Exclusion Criteria:

* Cognitive impairment
* Incarceration
* Under 21 years of age
* Adult unable to consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Receipt of Clinical Cancer Preventive Services and Resolution of Social Determinants of Health Barriers | through study completion, an average of 18 months
  Patient Receipt of Clinical Cancer Preventive Services and Resolution of Social Determinants of Health (SDoH) Barriers is an adjusted, composite proportion of items completed/resolved in 2 domains: (1) USPSTF recommended cancer screenings, behavioral counseling, and immunizations; and (2) SDoH barriers resolved from those identified in the Accountable Health Communities Health-Related Social Needs (AHC HRSN) Screening Tool

SECONDARY OUTCOMES:
Timeliness of diagnostic resolution | through study completion, an average of 18 months
  Time from an abnormal screening result to diagnostic resolution
Timeliness of treatment initiation | through study completion, an average of 18 months
  Time from diagnostic resolution to initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Simon, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern, Chicago, Illinois, United States